CLINICAL TRIAL: NCT05142046
Title: Influence of Intraoperative Fluid Balance on the Incidence of Adverse Events in Pediatric Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Denis SCHMARTZ, Head, Department of Anesthesiology, Brugmann University Hospital
Other Study IDs: CHUB_PED_Liquids-Cardiac
Record Dates: First submitted 2021-11-08; First posted 2021-12-02 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Congenital Heart Disease in Children; Surgery; Fluid Overload
MeSH Terms: conditions — Edema | interventions — Water-Electrolyte Balance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric cardiac surgery: The group consists of all the children who undergo cardiac surgery in our institution from 2008 to 2018. The age limit was from birth to 16 years old.
  Interventions: Drug: Fluid balance

INTERVENTIONS:
Drug: Fluid balance — The intervention consists of classic and standardized anesthesia management of children undergoing cardiac surgery. All the data links to the fluid management will be extracted from the patient's chart in the intraoperative period as well as complications during the hospitalization in the postoperative period.

SUMMARY:
The intraoperative fluid balance during pediatric cardiac surgery is a very sensitive parameter given the low circulating volume and the complexity of anesthetic management but might be deleterious if inadequately managed. The hypothesis is that a highly positive intraoperative fluid balance increases the incidence of adverse events in the short and long term.

A retrospective observational study including all consecutive children admitted for cardiac surgery with cardiopulmonary bypass (CPB) from 2008 to 2018 in a tertiary children's hospital will be performed. A multivariate analysis will be carried out to study the effect of the fluid balance on the incidence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 0-16 years and
* Cardiac surgery with cardiopulmonary bypass and
* operated between 2008 and 2018 at the Queen Fabiola University Children's Hospital (tertiary children's hospital)

Exclusion Criteria:

* ASA (American Society of Anesthesiologists) score of 5
* Jehovah's Witnesses
* incomplete hospital record

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The cohort consist of every child aged between 0-16 years who undergoes CPB-assisted cardiac surgery from 2008 to 2018 in Queen Fabiola University Children's Hospital (tertiary children's hospital).
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Severe postoperative morbidity | From intervention until 28 days postoperatively
  Severe postoperative morbidity will be characterized as the presence of two or more of the following situations: respiratory failure, prolonged inotropic support, or renal failure. Respiratory failure will be defined as the requirement for mechanical ventilation for >82 hours at any time from Pediatric Intensive Care Unit admission to the time of tracheal extubation.
  Prolonged inotropic support will be characterized as hemodynamic support by continuous vasoactive drug infusion for >48 hours postoperatively (excluding dopamine or dobutamine ≤5 μg/kg/min). Renal failure will be characterized as the worst estimated postoperative creatinine clearance (eCCr) value showing a ≥75% reduction compared with the preoperative baseline eCCr.

SECONDARY OUTCOMES:
Incidence of new Neurological deficits | From intervention until 28 days postoperatively
  Neurological deficit will be characterized as a transient or permanent functional abnormality in a body region due to a reduction of brain function. The measurement will be the incidence of ischemic stroke, hemorrhagic stroke and cognitive dysfunctions.
Incidence of new infections | From intervention until 28 days postoperatively
  Infection will be characterized as the need for antibiotics other than the usual anti-staphylococcal prophylaxis initiated by the attending intensive care physician for a suspected or proven infection caused by any pathogen or for a clinical syndrome associated with a high probability of infection. Measurement will be the number of patients with new infections corresponding to this definition.
Duration of mechanical ventilation | From intervention until 28 days postoperatively
  Delay between the end of the operation and the extubation of the patient.
PICU and hospital length of stay | From intervention until 28 days postoperatively
  Delay between the end of the operation and the exit of the patient of the Pediatric Intensive care Unit and the delay between the end of the operation and the exit of the institution.

CONTACTS AND LOCATIONS:
Overall Officials: Denis Schmartz, MD, Principal Investigator — Brugmann University Hospital & HUDERF
Locations (1):
- Hôpital Universitaire des Enfants Reine Fabiola, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Szekely A, Sapi E, Kiraly L, Szatmari A, Dinya E. Intraoperative and postoperative risk factors for prolonged mechanical ventilation after pediatric cardiac surgery. Paediatr Anaesth. 2006 Nov;16(11):1166-75. doi: 10.1111/j.1460-9592.2006.01957.x. PMID 17040306
- [Background] Agarwal HS, Wolfram KB, Saville BR, Donahue BS, Bichell DP. Postoperative complications and association with outcomes in pediatric cardiac surgery. J Thorac Cardiovasc Surg. 2014 Aug;148(2):609-16.e1. doi: 10.1016/j.jtcvs.2013.10.031. Epub 2013 Nov 23. PMID 24280709
- [Background] Lex DJ, Toth R, Czobor NR, Alexander SI, Breuer T, Sapi E, Szatmari A, Szekely E, Gal J, Szekely A. Fluid Overload Is Associated With Higher Mortality and Morbidity in Pediatric Patients Undergoing Cardiac Surgery. Pediatr Crit Care Med. 2016 Apr;17(4):307-14. doi: 10.1097/PCC.0000000000000659. PMID 26914622
- [Background] Stein A, de Souza LV, Belettini CR, Menegazzo WR, Viegas JR, Costa Pereira EM, Eick R, Araujo L, Consolim-Colombo F, Irigoyen MC. Fluid overload and changes in serum creatinine after cardiac surgery: predictors of mortality and longer intensive care stay. A prospective cohort study. Crit Care. 2012 May 31;16(3):R99. doi: 10.1186/cc11368. PMID 22651844
- [Background] Holte K, Sharrock NE, Kehlet H. Pathophysiology and clinical implications of perioperative fluid excess. Br J Anaesth. 2002 Oct;89(4):622-32. doi: 10.1093/bja/aef220. No abstract available. PMID 12393365
- [Background] Seguin J, Albright B, Vertullo L, Lai P, Dancea A, Bernier PL, Tchervenkov CI, Calaritis C, Drullinsky D, Gottesman R, Zappitelli M. Extent, risk factors, and outcome of fluid overload after pediatric heart surgery*. Crit Care Med. 2014 Dec;42(12):2591-9. doi: 10.1097/CCM.0000000000000517. PMID 25072753